CLINICAL TRIAL: NCT03298087
Title: Systemic and Tumor-Directed Therapy for Oligometastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONCA-013-16F
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Newly Diagnosed Oligometastatic Prostate Cancer
Keywords: oligometastatic; SBRT; abiraterone; apalutamide
MeSH Terms: interventions — Radiosurgery; Leuprolide; apalutamide; abiraterone; Abiraterone Acetate

STUDY DESIGN:
Intervention Model Description: Single arm Phase II clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Radical prostatectomy (and post-operative fractionated radiotherapy for pT=3a, pN1, or positive margins), metastasis directed SBRT, and complete ADT with LHRH analog leuprolide, abiraterone acetate with prednisone, and apalutamide (ARN-509) for a total of six months of systemic therapy.
  Interventions: Procedure: radical prostatectomy; Radiation: stereotactic body radiotherapy; Drug: Leuprolide; Drug: apalutamide; Drug: abiraterone

INTERVENTIONS:
Procedure: radical prostatectomy — surgical removal of the prostate
Radiation: stereotactic body radiotherapy — Highly targeted radiation
  Other Names: SBRT
Drug: Leuprolide — Lowers serum testosterone
  Other Names: ADT
Drug: apalutamide — antiandrogen
  Other Names: ARN-509
Drug: abiraterone — Inhibits androgen synthesis
  Other Names: zytiga

SUMMARY:
This is a trial for patients with newly diagnosed metastatic prostate cancer with 5 or fewer sites of metastases. The trial involves surgery (removal of the prostate) or radiation to the prostate, six months of hormone therapy, and stereotactic body radiotherapy to the sites of metastasis.

DETAILED DESCRIPTION:
This is a single arm Phase II clinical trial in patients with newly diagnosed M1a,b prostate cancer and 1-5 radiographically visible metastases treated with radical prostatectomy (and post-operative fractionated radiotherapy for pT 3a, pN1, or positive margins) or radiation to the prostate, metastasis directed SBRT, and complete ADT with LHRH analog leuprolide, abiraterone acetate with prednisone, and apalutamide (ARN-509) for a total of six months of systemic therapy. The primary endpoint of our study is the percent of patients achieving a serum PSA of <0.05 ng/mL six months after recovery of serum testosterone (for patients undergoing radical prostatectomy) or PSA <nadir+2 (for patients undergoing prostate radiation).

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy confirmed diagnosis of prostate adenocarcinoma (primary small cell carcinoma of the prostate is not allowed, however adenocarcinoma with neuroendocrine differentiation is allowed)
2. Age 18
3. Presence of 1-5 visible metastases (by NaF PET-CT or PSMA PET-CT including diagnostic CT of the chest, abdomen, and pelvis)

   1. At least one metastasis must be M1a-b
   2. Visceral metastases are not allowed
   3. Patients may have any number of pelvic nodal metastases (but largest must be <2 cm)
   4. Metastases must be amenable to treatment with SBRT
   5. Biopsy of one metastasis must be attempted, unless unsafe to perform. If biopsy is not diagnostic, or unsafe to perform, then a secondary imaging modality (for example, MRI) must also be consistent with metastatic disease (unless PSMA PET-CT was used as initial staging).
4. Patient must be fit to undergo radical prostatectomy, SBRT to all visible sites of metastases, ADT,
5. Total testosterone >200 ng/dL prior to ADT (optimal time to measure total testosterone is between 8 and 9 am)
6. Adequate performance status (ECOG 0-1)
7. Clinical laboratory values at screening:

   1. Hemoglobin 9.0 g/dL, independent of transfusion and/or growth factors within 3 months prior to randomization
   2. Platelet count 100,000 x 109/ L independent of transfusion and/or growth factors within 3 months prior to randomization
   3. Serum albumin 3.0 g/dL
   4. GFR 45 mL/min
   5. Serum potassium 3.5 mmol/L
   6. Serum total bilirubin 1.5 ULN (Note: In subjects with Gilbert's syndrome, if total bilirubin is >1.5 ULN, measure direct and indirect bilirubin and if direct bilirubin is 1.5 ULN, subject may be eligible)
   7. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <2.5 ULN
8. Medications known to lower the seizure threshold (see list under prohibited medications) must be discontinued or substituted at least 4 weeks prior to study entry.

Exclusion Criteria:

1. Any evidence of spinal cord compression (radiological or clinical)
2. Prior pelvic malignancy
3. Prior pelvic radiation
4. Concurrent malignancy aside from superficial skin cancers or superficial bladder tumors
5. Inability to undergo prostatectomy, radiotherapy, or ADT
6. Primary small cell carcinoma of the prostate (prostate adenocarcinoma with neuroendocrine differentiation is allowed)
7. Inflammatory bowel disease or active collagen vascular disease
8. History of any of the following:

   1. Seizure or known condition that may pre-dispose to seizure (e.g. prior stroke within 1year to randomization, brain arteriovenous malformation, Schwannoma, meningioma, or other benign CNS or meningeal disease which may require treatment with surgery or radiation therapy)
   2. Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to randomization
9. Current evidence of any of the following:

   1. Uncontrolled hypertension
   2. Gastrointestinal disorder affecting absorption
   3. Active infection (eg, human immunodeficiency virus [HIV] or viral hepatitis)
   4. Any chronic medical condition requiring a higher dose of corticosteroid than 10 mg prednisone/prednisolone once daily
   5. Any condition that in the opinion of the investigator would preclude participation in this study
   6. Concomitant strong CYP3A4 inducers. (If a strong CYP3A4 inducer must be co-administered, abiraterone acetate dose frequency will be adjusted).
   7. Treatment with CYP2D6 substrates that have a narrow therapeutic index. If an alternative treatment cannot be used, a dose reduction of the CYP2D6 substrate may be considered.
   8. Baseline severe hepatic impairment (ChildPugh Class B & C)
10. Presence of visceral metastases (i.e., stage M1c)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer only affects males.
Enrollment: 28 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas George Nickols, MD PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (3):
- United States (3):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parikh NR, Huiza C, Patel JS, Tsai S, Kalpage N, Thein M, Pitcher S, Lee SP, Inouye WS, Jordan ML, Sanati H, Jafari L, Bennett CJ, Gin GE, Kishan AU, Reiter RE, Lewis M, Sadeghi A, Aronson WJ, Garraway IP, Rettig MB, Nickols NG. Systemic and tumor-directed therapy for oligometastatic prostate cancer: study protocol for a phase II trial for veterans with de novo oligometastatic disease. BMC Cancer. 2019 Apr 1;19(1):291. doi: 10.1186/s12885-019-5496-5. PMID 30935383

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Arm
Started | 28
Completed | 24
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Arm
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 69 [62 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With PSA<0.05ng/mL (Radical Prostatectomy) or PSA <Nadir+2ng/mL (Prostate Radiation)
Description: PSA is a biomarker for disease burden in prostate adenocarcinoma and offers a non-invasive and sensitive assessment of disease control after treatment in the vast majority of patients.
Time Frame: 6 months after recovery of testosterone
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 24
Participants | 20

2. Secondary Outcome: Time to Biochemical Progression
Description: biochemical, radiographic, or clinical
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 24
months | NA [NA to NA] — Median and 95% Confidence Interval would not be reached because there were only three biochemical progressions.

3. Secondary Outcome: Time to Radiographic Progression
Description: per PCWG3 criteria
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 24
months | NA [NA to NA] — Median and 95% Confidence Interval would not be reached because there were only three radiographic progressions.

4. Secondary Outcome: Time to Initiation of Additional Antineoplastic Therapy
Description: antineoplastic therapy includes any systemic or focal anti-prostate cancer therapy
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 24
months | NA [NA to NA] — Median and 95% Confidence Interval would not be reached because there were only three who had addition antineoplastic therapy initiated.

5. Secondary Outcome: Prostate Cancer Specific Survival
Description: Prostate cancer specific survival
Time Frame: up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 24
percentage of participants | 100

6. Secondary Outcome: Patient Reported Outcomes as Assessed by Functional Assessment of Cancer Therapy - Prostate (FACT-P) Scale - Patient Questionnaire
Description: This uses the Functional Assessment of Cancer Therapy - Prostate (FACT-P) questionnaire. It assesses patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by 12 site specific items to assess for prostate related symptoms. Items are rated on a 0 to 4 Likert type scale and combined to produce sub-scores that are summed into a total FACT-P score, the higher the score, the better the quality of life. Range from 0-150 . Data was aggregated per patient and over time. Data represented here are the mean scores and 95% confidence intervals of the participants who filled out the questionnaire (15/24 completed through 18 months, 12/24 completed through 21 months).
Time Frame: Every 3 months up to a total of 21 months
Population: We could only analyze patients who agreed to fill out the questionnaires.
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Experimental Arm
Number analyzed (Participants) | 24
Score on a Scale
  Month 0: number analyzed (Participants) | 15
  Month 0 | 118 [108 to 129]
  Month 3: number analyzed (Participants) | 14
  Month 3 | 112 [103 to 122]
  Month 6: number analyzed (Participants) | 14
  Month 6 | 115 [106 to 124]
  Month 9: number analyzed (Participants) | 15
  Month 9 | 119 [107 to 131]
  Month 12: number analyzed (Participants) | 13
  Month 12 | 120 [110 to 131]
  Month 15: number analyzed (Participants) | 13
  Month 15 | 120 [108 to 131]
  Month 18: number analyzed (Participants) | 15
  Month 18 | 122 [112 to 133]
  Month 21: number analyzed (Participants) | 12
  Month 21 | 113 [100 to 127]

7. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by Physician Using CTCAE v4.0 Criteria
Description: CTCAE v4 criteria are a set of criteria for the standardized classification of adverse effects cancer therapy. The CTCAE system is a product of the US National Cancer Institute. The criteria are assessed by physician. The grades range from 0 to 5 (higher is worse). Data will be aggregated per patient and over time and classified by organ system (e.g., genitourinary, gastrointestinal, etc).
Time Frame: up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 24
Participants
  Grade 2 | 19
  Grade 3 | 2
  Grade 4 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 60 months after start date.
Description: Functional Assessment of Cancer Therapy-Prostate (FACT-P) was recorded every 3 months from baseline to a max of 21 months.
Arm/Group | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 1/28
Other Adverse Events (participants affected / at risk) | 21/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=28)
hypokalemia (Blood and lymphatic system disorders) | 1 (1) — 1 participant had grade 4 hypokalemia.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=28)
hypertension (Cardiac disorders) | 7 (7) — 7 participants had grade 2 hypertension
hypertension (Cardiac disorders) | 1 (1) — 1 participant had grade 3 hypertension
transaminitis (Hepatobiliary disorders) | 2 (2) — 2 participants had grade 2 transaminitis
rash (Skin and subcutaneous tissue disorders) | 3 (3) — 3 participants had grade 2 rash
concentration impairment (Nervous system disorders) | 1 (1) — 1 participant had grade 2 concentration impairment
incontinence (Renal and urinary disorders) | 7 (7) — 7 participants had grade 2 incontinence
cystitis (Renal and urinary disorders) | 1 (1) — 1 participant had grade 2 cystitis
urinary urgency (Renal and urinary disorders) | 2 (2) — 2 participants had grade 2 urinary urgency
urinary flow requiring tamsulosin (Renal and urinary disorders) | 4 (4) — 4 participants had grade 2 urinary flow requiring tamsulosin
rectal proctitis (Gastrointestinal disorders) | 1 (1) — 1 participant had grade 3 rectal proctitis

LIMITATIONS AND CAVEATS:
Limitations include the moderate sample size and the lack of a control arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT03298087/Prot_SAP_000.pdf